CLINICAL TRIAL: NCT04040075
Title: Open-label Switch Study From a Regimen of Elvitegravir/Tenofovir Alafenamide/Emtricitabine/Cobicistat and Darunavir, to a FDC of Bictegravir/Tenofovir Alafenamide/Emtricitabine in Virologically Suppressed HIV-l Subjects Known to Have an 184 V/I Mutation
Brief Title: Testing the Safety and Efficacy of Commercial Drug Biktarvy in Subjects Known to Have the 184 Resistance Mutation to a Component in Biktarvy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to complete enrollment goals due to unanticipated factors of screen failures, covid pandemic, and continued staffing and enrollment difficulties
Sponsor: Southampton Healthcare, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 184 Resistance Study
Record Dates: First submitted 2019-07-11; First posted 2019-07-31 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: subjects under current treatment for HIV with the I84 I/V Mutation Resistance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label (Other): Open label Biktarvy to establish suppression of HIV 1 with 184 V/I Resistance Mutation
  Interventions: Drug: Biktarvy Tab

INTERVENTIONS:
Drug: Biktarvy Tab — Antiretroviral drug

SUMMARY:
An Open-Label Study to Evaluate Switching from a Regimen of Elvitegravir/Tenofovir alafenamide/Emtricitabine/Cobicistat and Darunavir, to a Fixed-Dose Combination of Bictegravir/Tenofovir alafenamide/Emtricitabine in Virologically Suppressed HIV-1 Subjects who are known to have a I84 V/I Mutation

DETAILED DESCRIPTION:
An Open-Label Study to Evaluate Switching from a Regimen of Elvitegravir/Tenofovir alafenamide/Emtricitabine/Cobicistat and Darunavir, to a Fixed-Dose Combination of Bictegravir/Tenofovir alafenamide/Emtricitabine in Virologically Suppressed HIV-1 Subjects who are known to have a I84 V/I Mutation

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign a written informed consent which must be obtained prior to initiation of study procedures.
* Age equal to or greater than 18 years.
* Currently receiving an ARV regimen of EVG/F/TAF +DRV greater than six month.
* Documented plasma HIV - 1 RNA less than 50 copies/ml during the treatment with Elvitegravir/F/TAF for a minimum of 12 months prior to screening, on two separate determinations, with one determination within 3 months prior to screening.
* Have a documented 184 V/I resistant mutation.
* HIV-1 RNA levels < 50 copies per ml at screening.
* Estimated GFR >than or equal to 30 mls/min.
* AST and ALT equal to or less than 5 times upper limit of normal.
* Total bilirubin less than or equal to 1.5 mg/dl or normal direct bilirubin.
* Adequate hematologic function (absolute neutrophil count equal to or greater than 750/mm to the third, platelets equal to or greater than 50,000/mm to the third, Hemoglobin equal to or greater than 8.5 g/dl).
* Persons of child bearing potential must have negative serum pregnancy test at screening.
* Male participants and persons of child bearing potential who engage in heterosexual intercourse must agree to use our protocol specified methods of contraception.
* Female participants must agree to refrain from egg donation from first dose of FDC of B/F/TAF and throughout the study.
* Male participants must agree to refrain from sperm donation from first dose until at least 30 days after last dose of drug.
* Life expectancy equal to or greater than one year.

Exclusion Criteria:

* No desire to switch from current antiretroviral treatment.
* Any previous use of B/F/TAF.
* Any opportunistic illness indicative of stage 3 HIV diagnosed within 30 days prior to screening.
* Malignancy within 5 years of screening other than cutaneous Kaposi's sarcoma, completed resected non melanoma skin cancer, basal cell carcinoma, or noninvasive cutaneous squamous carcinoma, or completed resected carcinoma in situ of the cervix or anus. A prior malignancy treated with curative therapy and for which there has been no evidence of disease for at least 5 years prior to screening.
* Known hypersensitivity to FDC of B/F/TAF tablets their metabolites or formulation.
* No active treatment of Hepatitis C during the 48 weeks of the study.
* Females who are pregnant confirmed by serum pregnancy test.
* Females who are breast feeding.
* Suspected Biktarvy resistance mutations, except 184 V/I.
* Patients who need to take Dofetilide, Rifampin, Rifapentine, Rifabutin, phenobarbital, phenytoin, carbamazepine, oxcarbazepine, and antiretrovirals not part of the study and St. John's Wart during.
* Acute Hepatitis in the 30 days prior to screening.
* Active tuberculosis infection.
* Current alcohol or substance use judged by the investigator to potentially interfere with subject study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Test the safety and effectiveness of the drug Biktarvy in subjects known to have the 184 V/I resistance mutation. | In 48 week study
  Pure Virologic Response (PVR) with HIV-1 RNA < 50 copies/mL at week 12.

SECONDARY OUTCOMES:
Test the safety and effectiveness of the drug Biktarvy in subjects known to have the 184 V/I resistance mutation. | In 48 Week study
  Pure Virologic Response (PVR) with HIV-1 RNA < 50 copies/mL at week 24.
Test the safety and effectiveness of the drug Biktarvy in subjects known to have the 184 | 48 Weeks
  Pure Virologic Response (PVR) with HIV-1 RNA < 50 copies/mL at week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton Healthcare, Inc., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No